CLINICAL TRIAL: NCT03274908
Title: Real-world Clinical Study and Medical Machine Intelligence Study for Traditional Chinese Internal Medicine by Using Medical Big Data and Artificial Intelligence Methods
Brief Title: Real-world Clinical Study and Medical Machine Intelligence Study for Traditional Chinese Internal Medicine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Collaborators: Huashan Hospital (Other); Puer Hospital of Chinese Medicine (Unknown); Dangyang Hospital of Chinese Medicine (Unknown); Changde Hospital affiliated to Hunan University of Chinese Medicine (Unknown); Ruikang Hospital affiliated to Guanxi University of Chinese Medicine (Unknown); Jining First People's Hospital (Other); People's Hospital of Dangyang (Other)
Responsible Party: Principal Investigator, Zihui Tang, Principal Investigator, Huashan Hospital
Other Study IDs: 20170906
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Internal Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group
  Interventions: Other: regular medical treatment

INTERVENTIONS:
Other: regular medical treatment — regular medical treatment

SUMMARY:
This real-world study aimed at 1. exploring the relationships of traditional Chinese medicine (TCM) syndrome and internal diseases, 2. investigating the relationships of TCM treatment and internal diseases, and 3. creating medical machine intelligence to help internal physician in clinical practice. Big data methods and artificial intelligence algorithms are used to assess the associations based on electronic case files of patients.

ELIGIBILITY:
Inclusion Criteria:

* all patient records of internal medicine in hospital

Exclusion Criteria:

* subjects with major missing data

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients of internal medicine in hospital to include hospital of Chinese medicine and morden hospital in China
Sampling Method: Probability Sample
Enrollment: 2000000 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
internal diseases | 10 years
  all of internal diseases

CONTACTS AND LOCATIONS:
Locations (1):
- Huasha Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu J, Xu F, Mohammadtursun N, Lv Y, Tang Z, Dong J. The Analysis of Constitutions of Traditional Chinese Medicine in Relation to Cerebral Infarction in a Chinese Sample. J Altern Complement Med. 2018 May;24(5):458-462. doi: 10.1089/acm.2017.0027. Epub 2017 Aug 18. PMID 28820606
- [Background] Li X, Lei T, Tang Z, Dong J. Analyzing the association between fish consumption and osteoporosis in a sample of Chinese men. J Health Popul Nutr. 2017 Apr 19;36(1):13. doi: 10.1186/s41043-017-0088-y. PMID 28424092
- [Derived] Geng W, Qin X, Yang T, Cong Z, Wang Z, Kong Q, Tang Z, Jiang L. Model-Based Reasoning of Clinical Diagnosis in Integrative Medicine: Real-World Methodological Study of Electronic Medical Records and Natural Language Processing Methods. JMIR Med Inform. 2020 Dec 21;8(12):e23082. doi: 10.2196/23082. PMID 33346740